CLINICAL TRIAL: NCT06455800
Title: Long Term Outcome of Severe Lung Disease in Childhood
Brief Title: Severe Lung Disease in Childhood
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HCA-Lung
Record Dates: First submitted 2024-05-14; First posted 2024-06-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Lung Disease Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lung function measurements — Patients will once a year be monitored with different lung function methods

SUMMARY:
Only little information exists about the long term consequences of having severe lung disease in childhood. The patient population is heterogenous and the prognostic markers are few.

This observational study will investigate which parameters that can be used to predict the outcome of having severe lung disease in childhood.

DETAILED DESCRIPTION:
All patients aged 0-18 years at the HCA Childrens Hospital with a severe lung disease will prospectively be registered in a database.

At a yearly follow up, data from the patient record will be registered. Informed consent from the patients and/or their parents will be obtained. Registered data will include height, weight, results of lung function tests and imaging diagnostics.

The study will provide knowledge of the prognosis of different lung diseases and how to monitor lung function in children.

ELIGIBILITY:
Inclusion Criteria: severe lung disease -

Exclusion Criteria: no informed consent

-

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with severe chronic lung desease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
FEV1 | 18 years
  liter
FVC | 18 years
  liter
Lung Clearance Index (LCI) | 18 years
  number

SECONDARY OUTCOMES:
height | 18 years
  meters

CONTACTS AND LOCATIONS:
Overall Officials: Josefine Gradman, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Hans Christian Andersen Children's Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No